CLINICAL TRIAL: NCT05059639
Title: Exploring the Role of Almonds in Enhancing Immune Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Mark Kern, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-06-18
Record Dates: First submitted 2021-03-05; First posted 2021-09-28 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Immune Health
Keywords: Almonds

STUDY DESIGN:
Intervention Model Description: forty-eight overweight/non-obese (BMI=24-30) adult (ages 40-65 years) men (n=24) and women (n=24) will be recruited to participate. A randomized, parallel-arm design will be utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Almond (2 ounces) (Experimental): Consume 2 ounces almond daily for 8 weeks
  Interventions: Other: Almond
- Pretzel (Active Comparator): Consume comparative amount of pretzel for 8 weeks
  Interventions: Other: Pretzel

INTERVENTIONS:
Other: Almond — Consume 2 ounces of almond daily for 8 weeks
  Arms: Almond (2 ounces)
Other: Pretzel — Consume comparative amount of pretzel daily for 8 weeks
  Arms: Pretzel

SUMMARY:
The COVID-19 pandemic highlights the importance of good nutritional status for immune strength and for reducing comorbidities that increase morbidity and mortality of infections. The major aim of this study is test if almond consumption can improve immune function.

DETAILED DESCRIPTION:
Investigators will conduct an 8-week parallel-arm trial of 48 overweight/non-obese (BMI=24-30) adult (aged 40-65 years) men (n=24) and women (n=24) who will be randomly assigned to consume daily isoenergetic portions of almonds or a common snack (pretzels).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 40-65 y
* Body mass index (BMI) 24-30 kg/m.2

Exclusion Criteria:

* Not willing to stop taking multivitamins, and supplements (with the exception of vitamin D and calcium), for 30 days prior to or during study participation, if currently taking these.
* Almond allergies
* Alcohol consumption >2 drinks per day.
* Smoking or using nicotine containing products in the last 6 months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
change in Natural Killer Function | Baseline, after 8 weeks
  The ability of peripheral blood mononuclear cells to bind and kill leukemia cells will be measured at baseline and at week-8 of the diet intervention using flowcytometry by assessing the concentration of natural killer cells.

SECONDARY OUTCOMES:
change in Cytokines | Baseline, after 8 weeks
  Peripheral blood will be analyzed at baseline and week-8 of diet intervention for cytokines including IL1, IL-6 and TNF alpha concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hooshmand, PhD, RD, Study Director — San Diego State University
Locations (1):
- Mark Kern, PhD, RD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No